CLINICAL TRIAL: NCT07203287
Title: Risk of Acute Complications With Rocuronium vs Cisatracurium in Patients With Chronic Kidney Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-0406
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Post Operative Pulmonary Complications; Neuromuscular Blockade; General Anesthesia
MeSH Terms: interventions — Rocuronium; cisatracurium; Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rocuronium and Sugammadex (RS) Group (Active Comparator): The participants will be given rocuronium and sugammadex as part of one of the standard regimens of neuromuscular blockade and reversal.
  Interventions: Drug: Rocuronium; Drug: Sugammadex
- Cisatracurium and Neostigmine (CN) Group (Active Comparator): The participants will be given cisatracurium and neostigmine as part of one of the standard regimens of neuromuscular blockade and reversal.
  Interventions: Drug: Cisatracurium; Drug: Neostigmine

INTERVENTIONS:
Drug: Rocuronium — Will be assessing neuromuscular blockade with rocuronium and reversal with sugammadex
  Arms: Rocuronium and Sugammadex (RS) Group
Drug: Cisatracurium — Will be assessing neuromuscular blockade with neostigmine and reversal with neostigmine
  Arms: Cisatracurium and Neostigmine (CN) Group
Drug: Sugammadex — Will be assessing neuromuscular blockade with rocuronium and reversal with sugammadex
  Arms: Rocuronium and Sugammadex (RS) Group
Drug: Neostigmine — Will be assessing neuromuscular blockade with neostigmine and reversal with neostigmine
  Arms: Cisatracurium and Neostigmine (CN) Group

SUMMARY:
The purpose of the study is to determine which combination of neuromuscular blocking agent and reversal agent is safer to use during anesthesia for patients with chronic kidney disease. The main question it aims to answer is

"The use of Cisatracurium with neostigmine leads to less post-operative pulmonary complications than Rocuronium with sugammadex."

DETAILED DESCRIPTION:
Participants will be randomized into one of the two groups (Group 1-Given rocuronium and sugammadex as part of one of the standard regimens of neuromuscular blockade and reversal or Group 2-Given cisatracurium and neostigmine as part of one of the standard regimens of neuromuscular blockade and reversal).

Both of which are current standard of care practices. Appropriate reversal will be performed and documented, and the patient will go to the recovery room or intensive care unit as planned preoperatively. The patients will be assessed postoperatively for up to 7 days for any signs of respiratory complications, including but not limited to:

1. Atelectesis
2. Hypoxia
3. Respiratory distress/failure
4. Pneumonia
5. Pneumothrax

ELIGIBILITY:
Inclusion Criteria:

* The subject is able and willing to provide and sign informed consent
* The subject must be between 18 and 80 years of age
* The subject should have chronic kidney disease as defined by glomerular filtration rate
* The surgery must require general anesthesia with endotracheal intubation and neuromuscular blockade

Exclusion Criteria:

* Any patient under the age of 18
* Any patient over the age of 80
* Any patient with end stage renal disease
* Any patient requiring dialysis
* Patients presenting for Renal Transplantation
* Pregnant Female
* Any patient in the correctional system
* Urgent or Emergent procedure
* The surgery requires intubation post-operatively
* Documented allergy to Rocuronium, Sugammadex, Cisatracurium or Neostigmine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-26 (Estimated)

PRIMARY OUTCOMES:
Post Operative Pulmonary Complications (PPCs) | 7 days
  PPCs will be scored using a grading scale where 0 = no complication, 1 = mild, 2 = moderate, and 3 = severe complication, with 0 as the minimum score and 3 as the maximum score.

SECONDARY OUTCOMES:
Hospital Length of Stay | 7 days
  The total number of days the participant spent in the hospital.
Post Anesthesia Care Unit (PACU) length of stay | 7 days
  The total number of days the patient spent in the PACU.
Number of patients with cardiac instability | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Arango, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No